CLINICAL TRIAL: NCT04053283
Title: A Multicentre, Open-label, Non-randomised First in Human Study of NG-641, a Tumour Selective Transgene Expressing Adenoviral Vector, in Patients With Metastatic or Advanced Epithelial Tumours (STAR)
Brief Title: First in Human Study With NG-641, a Tumour Selective Transgene Expressing Adenoviral Vector
Acronym: STAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NG-641-01
Record Dates: First submitted 2019-08-09; First posted 2019-08-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Cancer; Epithelial Tumor
Keywords: metastatic; epithelial; virus; advanced; PsiOxus
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous (Experimental): Phase 1a dose escalation: one cycle of treatment.
  Phase 1a dose optimisation: up to 8 cycles of treatment
  Interventions: Biological: NG-641

INTERVENTIONS:
Biological: NG-641 — NG-641 is a replication competent adenoviral vector producing a bispecific T cell activator (TAc) targeting fibroblast activation protein (FAP) plus immune enhancer genes CXCL9/CXCL10/IFNa2. This can lead to killing of tumor cells and stimulation of immunity against the tumor cells.

SUMMARY:
To characterise the safety and tolerability of NG-641 in patients with metastatic or advanced epithelial tumours.

DETAILED DESCRIPTION:
To characterise the safety and tolerability of NG-641 in patients with metastatic or advanced epithelial tumours.

The Phase 1a part of the study is a dose-escalation and dose-optimization phase investigating NG-641 administration by intravenous (IV) infusion in a range of tumour types.

The Phase 1b part of the study will investigate the selected optimized multicycle dosing regimen as a monotherapy in up to three cohorts of patients with specific tumour types (Dose Expansion Cohorts A, B and C).

ELIGIBILITY:
Inclusion Criteria:

Phase 1a:

- Histologically or cytologically documented metastatic or advanced epithelial cancer that has relapsed from or is refractory to standard treatment, or for which no standard treatment is available

All patients

1. Provide written informed consent to participate
2. At least one measurable site of disease according to RECIST Version 1.1 criteria
3. Tumour accessible for biopsy, biopsy deemed safe by the Investigator, and patient willing to consent to tumour biopsies
4. Ability to comply with study procedures in the Investigator's opinion
5. Aged 18 years or over
6. ECOG performance status 0 or 1
7. Predicted life expectancy of 6 months or more
8. Adequate lung reserve
9. Adequate renal function
10. Adequate hepatic function
11. Adequate bone marrow function
12. Meeting reproductive status requirements

Exclusion Criteria:

1. Prior or planned allogenic or autologous bone marrow or organ transplantation
2. Splenectomy
3. Active infections requiring antibiotics, physician monitoring or systemic therapy within 1 week of the anticipated first dose of study drug, or recurrent fevers (>38.0˚C) associated with a clinical diagnosis of active infection
4. Treatment with the antiviral agents: ribavirin, adefovir, lamivudine, cidofovir or paxlovid within 10 days prior to the first dose of study treatment; or pegylated interferon in the 4 weeks before the first dose of study treatment
5. Known history of hepatitis B infection or known active hepatitis C infection. Known history of HIV infection
6. Patients who have active, known or suspected autoimmune disease that has required systemic therapy in the past 2 years, are immunocompromised in the opinion of the Investigator, or are receiving systemic immunosuppressive treatment
7. Treatment with any live, live-attenuated or COVID-19 vaccine in the 28 days before the first dose of NG-641
8. Treatment with any vaccine (including known non-adenoviral COVID-19 vaccines) in the 7 days before the first dose of NG-641
9. History of prior Grade 3-4 acute kidney injury or other clinically significant renal impairment
10. History of clinically significant interstitial lung disease or non-infectious pneumonitis
11. Lymphangitic carcinomatosis
12. Infectious or inflammatory bowel disease in the 3 months before the first dose of study treatment
13. Any known CTCAE Grade ≥2 coagulation abnormality/coagulopathy
14. Any clinically significant cardiovascular, peripheral vascular, cerebrovascular, or thromboembolic event in the 6 months before the first dose of study treatment
15. Grade 3 or 4 gastrointestinal bleeding All toxicities attributed to prior anti-cancer therapy (including radiation therapy) other than alopecia must have resolved to Grade 1 or baseline before the first dose of study treatment
16. Tumour location/extent considered by the Investigator to present a significant risk if tumour flare or necrosis were to occur
17. Known retinopathy, including retinal haemorrhages, cotton wool spots, papilloedema, optic neuropathy and retinal artery or vein obstruction
18. Active clinically severe depression
19. Use of following prior therapies

    * Enadenotucirev-based therapy, or a fibroblast activation protein (FAP) targeting agent anytime
    * Anti-cancer monoclonal antibody (mAb), immune checkpoint inhibitor, immune stimulatory treatment or other biological therapy in the 28 days prior to the first dose of study treatment (PD-1 / PD-L1 therapy permitted without a 'washout' phase)
    * Chemotherapy, targeted small molecule or other investigational drug in the 14 days or five half-lives (whichever is shorter) before the first dose of study treatment
    * Major surgery in the 28 days before the first dose of study treatment or radiation therapy in the 14 days before the first dose of study treatment
    * Bisphosphonate therapy or treatment with Receptor Activator of Nuclear factor Kappa-Β (RANK)-ligand inhibitors for metastatic bone disease is permitted
20. All toxicities attributed to prior anti-cancer therapy (including radiation therapy) other than alopecia must have resolved to Grade 1 or baseline before the first dose of study treatment
21. Known allergy/immune-related adverse reactions to NG-641 transgene or immune checkpoint inhibitor products or formulation; severe hypersensitivity to another monoclonal antibody
22. Known hypersensitivity to both cidofovir and valacyclovir
23. Other prior malignancy active within the previous 3 years (see protocol for exceptions)
24. Symptomatic brain metastases or any leptomeningeal metastases that are symptomatic and/or requires treatment
25. Any serious or uncontrolled medical disorder that, in the opinion of the Investigator or the Medical Monitor, may increase the risk associated with study participation or study treatment administration, impair the ability of the patient to receive protocol therapy or interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (safety and tolerability) in study NG-641 | End of study treatment visit
  Incidence of adverse events, adverse events meeting protocol-defined DLT criteria, adverse events leading to study treatment or study discontinuation, and adverse events resulting in death.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Southern California (USC) - Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA, Santa Barbara, California
  - Moffitt-Advent Health Clinical Research Unit, Celebration, Florida
  - Ochsner Medical Center (OMC) - The Gayle and Tom Benson Cancer Center, New Orleans, Louisiana
  - Washington University Medical School, St Louis, Missouri
  - MD Anderson, Houston, Texas

REFERENCES:
- [Derived] Khalil DN, Prieto Gonzalez-Albo I, Rosen L, Lillie T, Stacey A, Parfitt L, Soff GA. A tumor-selective adenoviral vector platform induces transient antiphospholipid antibodies, without increased risk of thrombosis, in phase 1 clinical studies. Invest New Drugs. 2023 Apr;41(2):317-323. doi: 10.1007/s10637-023-01345-8. Epub 2023 Mar 10. PMID 36897458